CLINICAL TRIAL: NCT01145001
Title: Contingency Management for Smoking Cessation in Adolescent Smokers - Phase IV, Enhancing a High School Based Smoking Cessation Program
Brief Title: Enhancing a High School Based Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 020718574; P50DA009241-17 (NIH)
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Nicotine Dependence
Keywords: smoking; adolescents; contingency management; nicotine replacement therapy
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Cognitive Behavioral Therapy; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active Nicotine Patch and Contingency Management (Active Comparator): Subjects in this group will receive Contingency Management and active nicotine patch
  Interventions: Behavioral: Cognitive Behavioural Therapy; Behavioral: Contingency Management; Drug: Nicotine Transdermal Patch
- Nicotine Patch with no Contingency Management (Active Comparator): Subjects in this group will receive active nicotine patch without contingency management for abstinence
  Interventions: Behavioral: Cognitive Behavioural Therapy; Drug: Nicotine Transdermal Patch
- Placebo patch and Contingency Management (Placebo Comparator): Subjects in this group will receive a placebo transdermal patch and contingency management
  Interventions: Behavioral: Cognitive Behavioural Therapy; Behavioral: Contingency Management
- Placebo Patch and no Contingency Management (Placebo Comparator): Subjects in this group will receive a placebo patch and will not receive contingency management
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Weekly CBT for all subjects
Behavioral: Contingency Management — incentives given for abstinence based on urine analysis
  Arms: Active Nicotine Patch and Contingency Management; Placebo patch and Contingency Management
Drug: Nicotine Transdermal Patch — 14mg ir 21mg doses based on weight and #cigs/day
  Other Names: Habitrol
  Arms: Active Nicotine Patch and Contingency Management; Nicotine Patch with no Contingency Management

SUMMARY:
The purpose of this study is to examine the the efficacy of adjunctive nicotine replacement therapy when used in combination with the contingency management (CM) + cognitive behavioral therapy intervention. Subjects will be randomly assigned to receive either a nicotine transdermal patch or a placebo patch as well as being randomly assigned to receive either CM or no CM; all subjects will receive cognitive behavioral therapy. We hypothesize that that subjects receiving both active nicotine patch and CM will have higher rates of abstinence from tobacco than subjects in the other groups.

ELIGIBILITY:
Inclusion Criteria:

* High School aged
* Desire to quit smoking
* Smoking >5 cigarettes per day
* Able to read and write in English

Exclusion Criteria:

* Current dependence on other substances
* Medical conditions that would contraindicate the use of a nicotine patch

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2009-11; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- CMHC, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Nicotine Patch and Contingency Management | Nicotine Patch With no Contingency Management | Placebo Patch and Contingency Management | Placebo Patch and no Contingency Management
Started | 36 | 37 | 44 | 37
Completed | 28 | 31 | 39 | 31
Not Completed | 8 | 6 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Nicotine Patch and Contingency Management | Nicotine Patch With no Contingency Management | Placebo Patch and Contingency Management | Placebo Patch and no Contingency Management | Total
Number analyzed (Participants) | 36 | 37 | 44 | 37 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 36 | 42 | 37 | 149
  Between 18 and 65 years | 2 | 1 | 2 | 0 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.53 (1.276) | 16.62 (1.233) | 16.66 (1.01) | 16.30 (1.151) | 16.53 (1.161)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 14 | 17 | 17 | 59
  Male | 25 | 23 | 27 | 20 | 95
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 44 | 37 | 154

OUTCOME MEASURES:

1. Primary Outcome: Abstinence Rates at the End of Treatment
Description: Our primary outcome will be point prevalence abstinence at the end of the treatment period defined as any self-report of cigarette use during the seven days prior to the last appointment confirmed by urine analysis.
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants not smoking
Arm/Group | Active Nicotine Patch and Contingency Management | Nicotine Patch With no Contingency Management | Placebo Patch and Contingency Management | Placebo Patch and no Contingency Management
Number analyzed (Participants) | 36 | 37 | 44 | 37
percentage of participants not smoking | 35.1 | 24.3 | 38.6 | 36.1

2. Secondary Outcome: Continuous Abstinence During Treatment
Description: We will also examine continuous abstinence during the six week treatment period by urine analysis each week.
Time Frame: 6 weeks
Population: this is the intent to treat group-all starters (not treatment completers)
Measure: Mean (Standard Deviation); unit: consecutive days of abstinence
Arm/Group | Active Nicotine Patch and Contingency Management | Nicotine Patch With no Contingency Management | Placebo Patch and Contingency Management | Placebo Patch and no Contingency Management
Number analyzed (Participants) | 42 | 34 | 35 | 32
consecutive days of abstinence | 26.1 (14.1) | 26.6 (13.7) | 29 (14.7) | 30 (13)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline through duration of treatment-6 weeks
Arm/Group | Active Nicotine Patch and Contingency Management | Nicotine Patch With no Contingency Management | Placebo Patch and Contingency Management | Placebo Patch and no Contingency Management
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/44 | 0/37
Other Adverse Events (participants affected / at risk) | 32/36 | 33/37 | 42/44 | 33/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Nicotine Patch and Contingency Management (N=36) | Nicotine Patch With no Contingency Management (N=37) | Placebo Patch and Contingency Management (N=44) | Placebo Patch and no Contingency Management (N=37)
Nausea (Gastrointestinal disorders) | 14 | 11 | 10 | 14
Vomiting (Gastrointestinal disorders) | 8 | 4 | 5 | 7
Abdominal Pain (Gastrointestinal disorders) | 9 | 7 | 7 | 11
Change in appetite (General disorders) | 20 | 20 | 25 | 22
Headache (General disorders) | 19 | 24 | 26 | 22
Dizziness (Nervous system disorders) | 6 | 11 | 9 | 14
Blurred vision (Eye disorders) | 6 | 3 | 5 | 8
Rapid Heartbeat (Cardiac disorders) | 5 | 6 | 8 | 7
Fatigue (General disorders) | 11 | 13 | 13 | 17
Nervousness (Social circumstances) | 17 | 16 | 14 | 14
Insomnia (General disorders) | 17 | 13 | 15 | 11
Sleepiness (General disorders) | 12 | 13 | 20 | 16
Itching (Skin and subcutaneous tissue disorders) | 14 | 16 | 11 | 11
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 5 | 4
VIvid Dreams (Psychiatric disorders) | 15 | 15 | 15 | 12
Sweating (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 14 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes